CLINICAL TRIAL: NCT00129493
Title: Group Visits to Improve Hypertension Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRH 01-173
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2009-05

CONDITIONS: Hypertension
Keywords: Practice guidelines; Hypertension; Primary health care; Patient-centered care; Healthcare quality; Office visits; Self-efficacy; Self care; Guideline adherence; Patient noncompliance
MeSH Terms: conditions — Hypertension; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Group medical visits

INTERVENTIONS:
Behavioral: Group medical visits — Our intervention aims to develop and implement a model of group medical visits in iterative steps, to evaluate whether group medical visits improve patient adherence to prescribed antihypertensive medications and improve BP control, and to assess patient, physician, and health care system factors involved in successfully making organizational changes to encompass group medical visits.

SUMMARY:
This study investigates group medical visits as a quality improvement strategy for hypertension. It studies group visits in which patients see their own primary care provider together with other patients who have hypertension. The group visits are intended to enhance the patient's self-efficacy for self-management of their chronic disease (hypertension).

DETAILED DESCRIPTION:
BACKGROUND Many veterans with hypertension have poorly controlled blood pressure (BP); new strategies for quality improvement are needed. A new model of care delivery, Group Medical Visits, holds promise as a means to improve blood pressure control by enhancing patients' self-efficacy for self-management of their chronic disease.

Objectives The overriding goal of this implementation project is to translate research findings about management of hypertension into practice and thereby to improve patient outcome, i.e., adequacy of control of BP, in patients with hypertension. Specific objectives are to develop and implement a model of group medical visits in iterative steps; to evaluate whether group medical visits improve patient adherence to prescribed antihypertensive medications and improve BP control; and to assess patient, physician, and health care system factors involved in successfully making organizational changes to encompass group medical visits.

Methods Study site: primary care clinics at VA Palo Alto. Study Design: staircase design with 2 steps of design/implementation/formative-evaluation/redesign with increasing numbers of participants, followed by a 3rd step evaluating the final model. Participants: primary care providers (MDs and RNPs) and their patients with hypertension. Participating primary care providers (PCPs) are randomly allocated 2:1 Group Visits (GV)intervention:control; patients of intervention PCPs are also randomly allocated 2:1, yielding 3 study arms (patients of GV-PCPs enrolled in GVs; patients of GV-PCPs not in GVs, and patients of non-GV-PCPs). This design allows for comparison between control patients of primary care providers conducting group visits with primary care providers who do not participate in the group medical appointment intervention. Intervention: group medical visits of patients with their own PCP. Group visits include both education and medical care components. Organizational component: tracking of organizational issues in establishing the program of group visits; interviews with key stakeholders to identify barriers and facilitators to implementing the new model of care. Outcome measures: patients' blood pressures (BPs), medication adherence, satisfaction, and health-related quality of life; PCP satisfaction; qualitative analysis of themes from interviews for patient, physician, and medical center factors involved in making organizational changes to encompass group visits.

Findings We exceeded the target enrollment for primary care providers (PCPs) with a total of 16 (11 intervention, 5 control). We enrolled 296 patients; 7 had incomplete baseline data leaving 289 patients: 145 allocated to GVs, 73 control patients of GV-PCPs, and 71 control patients of control PCPs. We have also enrolled an additional 12 staff members for interviews, including the one PCP who did not elect to participate. Study arm comparisons will not be made until the final data collection is complete. In formative evaluations we found that patient medical needs were met in the group setting and that both patients and PCPs were satisfied with the GV format. PCPs and patients have requested that the GVs continue after the study ends. Space for the GVs has been a major barrier particularly in light of ongoing construction in the clinic building.

Status We are now in Step 3 with plans to end the intervention phase at the end of March 2006 and complete final data collection soon thereafter.

Impact Group Medical visits are a new model of health care delivery that hold promise for improving patient access, patient and provider satisfaction, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Subjects include both health care professionals and their patients. The included health care professionals are primary care clinicians practicing at VA Palo Alto who have their own panels of patients for whom they provide primary care. Included patients are patients of these primary care clinicians; the patients must have a diagnosis of hypertension and at least one blood pressure in the previous year that was above guideline-target for that patient, and patient must be approved by the primary care clinician as suitable for a group medical visit.

Exclusion Criteria:

Primary care clinicians with very small patient panels (too small for recruitment of patients for group visits) ae excluded. Patients are excluded by their primary care clinician using clinical judgment; typical reasons for exclusion include terminal illness, dementia that would make patient unable to participate in group discussions. Because primary care clinicians located at main study site do not provide primary care to children, no children will be included in the sample.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-02; Primary Completion 2006-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure from baseline to endpoint (6, 12 or 18 months depending on how long patient is in study) and comparisons of study arms; change inmedication adherence from baseline to endpoint. Formative evaluation of the program. | 6, 12, 18 months

SECONDARY OUTCOMES:
Patient, provider and other staff satisfaction; organizational impact of the group visits program (health care system factors exploratory analyses of utilization)added value of visits beyond 12 months, qualitative data from interviews. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary K. Goldstein, MD MS, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts

REFERENCES:
- See also: Stanford Community Profiles of Faculty: principal investigator information — http://med.stanford.edu/profiles/Mary_Goldstein/